CLINICAL TRIAL: NCT06112600
Title: The Impact of Virtual Reality and Kaleidoscope Usage on Pain, Fear, and Anxiety in Children During Routine Vaccination: A Randomized Controlled Study
Brief Title: The Impact of Virtual Reality and Kaleidoscope in Children During Vaccination
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Ege University (Other)
Responsible Party: Principal Investigator, Merve Gümüş, Research Assistant Dr., Ege University
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Supportive Care
Other Study IDs: E-79593712-799
Record Dates: First submitted 2023-10-23; First posted 2023-11-01 (Actual); Last update posted 2023-11-01 (Actual); Status verified 2023-10

CONDITIONS: Pain; Pediatric Patient; Fear; Virtual Reality; Nursing Caries
MeSH Terms: conditions — Pain

STUDY DESIGN:
Intervention Model Description: This prospective, randomised controlled study
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (3):
- Control Group (No Intervention): No attention-diverting method was applied to the children in this group and routine vaccination was administered.
- Virtual Reality group (Experimental): The VR group received a VR application using the Oculus Quest 2 while being vaccinated.
  Interventions: Procedure: VR
- Kaleidoscope group (Experimental): In the Kaleidoscope group, children were given a kaleidoscope toy while being vaccinated.
  Interventions: Procedure: Kaleidoscope

INTERVENTIONS:
Procedure: VR — Virtual reality glasses were used as a distraction method for children during vaccination.
  Arms: Virtual Reality group
Procedure: Kaleidoscope — Kaleidoscope toys were used as a distraction method for children during vaccination.
  Arms: Kaleidoscope group

SUMMARY:
This study was designed to examine the effects of using virtual reality and kaleidoscope during routine vaccination in children aged 48 months on pain, fear, and anxiety. Children aged 48 months who were to receive the measles-mumps-rubella vaccine were randomized into three groups. Accordingly, the study sample consisted of a virtual reality group with 42 children, a kaleidoscope group with 42 children, and a control group with 42 children, totaling 126 children. Fear and pain were evaluated by both the researcher and the child before and after the procedure. Anxiety was assessed by the child after the procedure. The Wong Baker Faces Pain Rating Scale was used for pain, the Children's Fear Scale for fear, and the Child Anxiety Scale-State Version for anxiety.

ELIGIBILITY:
Inclusion Criteria:

* being 48 months
* being conscious (with the ability to communicate).

Exclusion Criteria:

* Having a physical and psychological condition that prevents them from wearing glasses to view VR;
* Having a visual problem
* Having mental or physical disabilities
* Taking any analgesics, sedatives, or anticonvulsants in the past 24 hours
* Having chronic or life-threatening disease
* Refusing the VR or kaleidoscope intervention during vaccine injection.

Ages: 48 Months to 48 Months | Sex: All | Healthy Volunteers: No
Age Groups: Child
Enrollment: 126 (Actual)
Dates: Start 2021-09-15 (Actual); Primary Completion 2023-05-30 (Actual); Study Completion 2023-06-30 (Actual)

PRIMARY OUTCOMES:
Procedural Pain | 1 year
  Just before vaccination, both the child and the researcher used the Wong-Baker Faces Scale. This scale uses in children aged 3 and older to rate pain severity. This numeric rating scale ranges from 0 to 10. Faces show emotions from smiling (0 = very happy/no pain) to crying (10 = hurts worst). The child can choose the face that best illustrates the physical pain.
Fear | 1 year
  Just before vaccination, both the child and the researcher used the Children's Fear Scale. The scale includes five drawn facial expressions ranging from a neutral expression (0=no anxiety) to a frightened face (4=severe anxiety) and has been validated for the Turkish population The scale allows for evaluations on a scale from 0 to 4.
Anxiety | 1 year
  Just before vaccination, both the child and the researcher used the Children's Anxiety Meter-State. It is drawn like a thermometer with a bulb at the bottom. It includes horizontal lines going up to the top (0-10). Children are asked to mark how feel "right now" to measure state anxiety. Higher values represent higher anxiety.

SECONDARY OUTCOMES:
Parental satisfaction | 1 year
  parental satisfaction scores measured with the 10-point Likert type scale. Minimum score is 0, maximum score is 10.

CONTACTS AND LOCATIONS:
Locations (1):
- Ege University, Izmir, Bornova, Turkey (Türkiye)